CLINICAL TRIAL: NCT01023763
Title: Can a Structured Training Program in Intravenous Treatment of Infections in Nursing Homes Lead to a Better Patient Trajectory and Reduced Hospital Admittance?
Brief Title: Intravenous Treatment in Nursing Homes
Acronym: 3IV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Morten Lindbaek, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/1584a
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Infections; Dehydration
Keywords: Nursing homes; Intravenous; Treatment; Patient trajectory; Hospital admissions
MeSH Terms: conditions — Infections; Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Nursing home residents who require intravenous fluids and intravenous antibiotics was treated as usual (hospital admissions for intravenous treatment).
  In control nursing homes that had not completed the training program (intervention period), nursing home residents who require intravenous fluids and intravenous antibiotics was treated as usual. The majority of these patients were admitted to hospital for intravenous treatment. A few nursing homes or nursing home departments had sufficient expertise and capacity to provide treatment locally.
- A training program in iv treatment (Other): A structured training program in intravenous treatment in nursing homes:
  Each of 30 participating nursing homes sequentially received theory and practical training in intravenous treatment. In nursing homes that had completed the training program (intervention period), and had sufficient expertise and capacity, nursing home residents in need of intravenous fluids or antibiotics were treated locally; otherwise they were hospitalized.
  Interventions: Other: A structured training program

INTERVENTIONS:
Other: A structured training program — A structured training program in nursing homes in the intravenous treatment of dehydration and infections.
  Arms: A training program in iv treatment

SUMMARY:
The primary objective for the project is to evaluate whether nursing home residents who require intravenous fluids and intravenous antibiotics, can be treated just as well or even better in the nursing home as in the hospital. In Vestfold, Norway, a structured training program in the intravenous treatment of dehydration and infections in nursing homes is planned. The 3IV study will evaluate if this leads to an equal or better patient trajectory and reduced hospital admittance.

DETAILED DESCRIPTION:
1. Can a structured training program in administration of intravenous fluids and antibiotics lead to a reduced number of admissions and days in hospitals among nursing home residents?
2. Can treatment with intravenous fluids or antibiotics in nursing homes provide an equally good or better patient trajectory compared to patients hospitalized for the same treatment? We will look at duration of symptoms, direct and indirect complications, and mortality rates.
3. Can treatment costs for the public health service be reduced when patients are treated with intravenous fluids and /or antibiotics in the nursing home instead of being admitted to the hospital?
4. Can treatment for dehydration and infections in the nursing home rather than in a hospital provide an equally or better satisfaction in patients, next of kin and staff?
5. How are difficult ethical issues handeld by medical staff at the nursing homes and the hospital when nursing home patients receive intravenous treatment?

ELIGIBILITY:
Inclusion Criteria:

* Nursing home residents in need of intravenous fluids or antibiotics

Exclusion Criteria:

* Patients who needs hospitalization due to either co-morbidity or seriousness of disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
All cause morbidity and mortality | Within 30 days after disease onset

SECONDARY OUTCOMES:
Number of admissions and days in hospitals among nursing home residents | Primarily within 30 days after disease onset
Patient trajectory | Primarily within 30 days after disease onset
Satisfaction in patients, next of kin and staff | Primarily within 30 days after disease onset

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klomstad K, Pedersen R, Forde R, Romoren M. Involvement in decisions about intravenous treatment for nursing home patients: nursing homes versus hospital wards. BMC Med Ethics. 2018 May 8;19(1):34. doi: 10.1186/s12910-018-0258-5. PMID 29739393
- [Derived] Nyborg G, Brekke M, Straand J, Gjelstad S, Romoren M. Potentially inappropriate medication use in nursing homes: an observational study using the NORGEP-NH criteria. BMC Geriatr. 2017 Sep 19;17(1):220. doi: 10.1186/s12877-017-0608-z. PMID 28927372